CLINICAL TRIAL: NCT03725696
Title: The Effect of Bariatric Surgery on Spermatogenesis
Status: Terminated | Type: Observational
Why Stopped: •Terminated: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Scott Lundy, Resident Physician, The Cleveland Clinic
Other Study IDs: IRB 16-721
Record Dates: First submitted 2018-10-24; First posted 2018-10-31 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Bariatric Surgery Candidate; Sexual Function and Fertility Disorders
MeSH Terms: interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients who are booked for RYGB gastric bypass surgery and enroll in the study will undergo semen analysis, sexual health questionnaire (IIEF survey), and a blood hormonal panel before and after surgery.
  Interventions: Diagnostic Test: Semen Analysis; Diagnostic Test: Hormonal panel; Procedure: RYGB Gastric Bypass; Diagnostic Test: IIEF Survey

INTERVENTIONS:
Diagnostic Test: Semen Analysis — Sperm counts will be determined by semen analysis.
Diagnostic Test: Hormonal panel — Blood test for LH, FSH, testosterone, and estradiol
Procedure: RYGB Gastric Bypass — Roux-en-Y Gastric Bypass
Diagnostic Test: IIEF Survey — International Index of Erectile Function is a validated 5-question survey examining sexual health in men

SUMMARY:
Little is known about the effects of weight loss surgery on male reproductive health. This study will investigate the effect of bariatric surgery on male infertility by evaluating sexual health, blood hormone levels, and semen parameters before and after roux-en-y bariatric surgery.

DETAILED DESCRIPTION:
Obesity is a worldwide epidemic that has numerous health consequences including male infertility. Prior studies have shown a variety of health benefits with bariatric surgery, including an improvement/resolution in diabetes and a significant improvement in serum testosterone levels. Based upon preliminary data from the literature, the investigators hypothesize that bariatric surgery is associated with a transient decrease followed by a robust long-term improvement in semen parameters including DNA fragmentation and oxidative stress. To test this hypothesis, the investigators propose a prospective observational study examining changes in hormone and semen parameters over the 12 months following Roux-en-Y gastric bypass surgery. The investigators will correlate these changes to weight loss, changes in subjective sexual function, and advanced semen parameters including DNA fragmentation. If successful, this study will conclusively identify a new modifiable cause for male infertility and suggest an additional medical indication for bariatric surgery in obese infertile men.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-55
* Undergoing Roux-en-Y bariatric surgery

Exclusion Criteria:

* History of undescended testes
* Prior scrotal surgery
* Known karyotypic abnormalities

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Men between the ages of 18 and 50 scheduled for bariatric surgery who meet the above enrollment criteria will be offered enrollment in the study at the time of their preoperative clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in sperm concentration | Baseline to 12 months
  Changes in sperm concentration on semen analysis

SECONDARY OUTCOMES:
Weight loss | Baseline to 12 months
  Change in weight following bariatric surgery
Changes in sexual health | Baseline to 12 months
  Change in International Index of Erectile Function (IIEF) score, a validated questionnaire with scores ranging from 1 (significant erectile dysfunction to 30 (no erectile dysfunction).
Changes in reproductive hormones | Baseline to 12 months
  Changes in FSH, LH, testosterone, and estrogen blood levels
Changes in seminal oxidative stress | Baseline to 12 months
  Changes in seminal reactive oxygen species
Changes in sperm morphology | Baseline to 12 months
  Changes in percent normal sperm morphology on semen analysis
Changes in seminal DNA fragmentation | Baseline to 12 months
  Changes in seminal DNA fragmentation rate on semen analysis

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lundy, MD PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No